CLINICAL TRIAL: NCT02597114
Title: An Extension Study of AGT-181-102 Evaluating Safety and Glycosaminoglycans (GAGs) in Adult Patients With Hurler-Scheie or Scheie Syndrome Who Have Completed 8-Weeks of Dosing With AGT-181 in Study AGT-181-102
Brief Title: Extension Study of AGT-181-102 to Evaluate Long Term Safety and Activity of AGT-181
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArmaGen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGT-181-103
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Mucopolysaccharidosis I
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — valanafusp alpha

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AGT-181 (Experimental): AGT-181 (fusion protein of anti-human insulin receptor monoclonal antibody and alpha-L-iduronidase) administered once weekly x 26 weeks at same dose level as subject received in core study
  Interventions: Drug: AGT-181

INTERVENTIONS:
Drug: AGT-181 — intravenous infusion over 3-4 hours
  Other Names: HIRMAb-IDUA; fusion protein of monoclonal antibody to human insulin receptor fused to alpha-L-iduronidase

SUMMARY:
AGT-181 is a fusion protein containing alpha-L-Iduronidase that is intended to deliver the enzyme peripherally and to the brain, when administered intravenously. This study is an extension of a safety and dose ranging study to obtain long term safety and exposure data, as well as information on the biological activity of the investigational drug

ELIGIBILITY:
Inclusion Criteria:

* Must have completed clinical trial AGT-181-102
* Voluntary written consent by patient or legally responsible representative
* All women of childbearing potential and sexually mature males must be advised to use a medically accepted method of contraception throughout the study.
* Negative pregnancy test (females)

Exclusion Criteria:

* Refusal to complete screening evaluations.
* Any medical condition or other circumstances that may significantly interfere with study compliance
* Patient is pregnant or lactating
* Clinically significant spinal cord compression, evidence of cervical instability.
* Subject developed clinically relevant hypersensitivity to AGT-181

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 104 weeks (2 years)

SECONDARY OUTCOMES:
changes in urinary or plasma glycosaminoglycans (GAGs) | 104 weeks (2 years)
change in liver size | 104 weeks (2 years)
change in spleen size | 104 weeks (2 years)
change in levels of heparan sulfate and dermatan sulfate in the cerebrospinal fluid | 104 weeks (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Rioux, MD PhD, Study Director — ArmaGen, Inc